CLINICAL TRIAL: NCT02451917
Title: Subcutaneous Insulin Glargine Versus NPH Insulin in Patients With Chronic Kidney Disease Stages III and IV: Randomized Controlled Trial.
Brief Title: Glargine Versus NPH in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENDONEFRO
Record Dates: First submitted 2014-08-25; First posted 2015-05-22 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
Keywords: Glargine insulin; Chronic Kidney Disease; CGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Insulin Glargine; Insulin, Isophane; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glargine insulin (Experimental): This is an open-label, randomized, two-way crossover study , one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of insulin glargine, regardless of the sequence were grouped as glargine.
  Interventions: Drug: Glargine insulin
- NPH insulin (Active Comparator): This is an open-label, randomized, two-way crossover study , one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin.
  At the end of the study, all data acquired during the use of NPH insulin, regardless of the sequence were grouped as NPH.
  Interventions: Drug: NPH insulin

INTERVENTIONS:
Drug: Glargine insulin — The initial insulin dose for those randomized to IGlar was 80% of the total daily NPH dose that was being discontinued. All of them had pre-prandial Regular insulin switched to Lispro insulin (Humalog™, Lilly, Brazil), at the same dose as in use previously. After 24 weeks, basal insulins were switched; in other words, individuals on IGlar in the first period switched to INPH, and the doses of pre-meal insulin were sustained
  Other Names: Lantus insulin ™, Sanofi-Aventis, Brazil
  Arms: Glargine insulin
Drug: NPH insulin — The same total daily NPH insulin dose was maintained for those randomized to INPH. All of them had pre-prandial Regular insulin (Humulin R™, Lilly, Brazil) switched to Lispro insulin (Humalog™, Lilly, Brazil), at the same dose as in use previously. . After 24 weeks, basal insulins were switched; in other words, individuals on NPH in the first period switched to glargine insulin, and the doses of pre-meal insulin were sustained.
  Other Names: Humulin N™, Lilly, Brazil
  Arms: NPH insulin

SUMMARY:
Chronic kidney disease (CKD) is one of the most common microvascular complications of diabetes mellitus, and it is the leading cause of end stage renal disease on developed countries. The CKD diagnosis and its progression require re-evaluation of hypoglycemic therapy and constant dosing adjustments, in order to optimize glycemic control and minimize its side effects. Long acting insulin analogs and its pharmacokinetics have not been studied through different stages of kidney disease and there is no consensus defining the appropriate dosing adjustment based on the glomerular filtration rate (GFR). This research project will compare the glycemic response to intensive insulin treatment with NPH insulin and basal insulin analog (insulin glargine) in type 2 diabetes (DM 2) patients with CKD stages 3 and 4. Patients and methods - Inclusion Criteria: DM 2 patients with CKD secondary to diabetic nephropathy and GFR of 15-59 ml/min/1.73m². Exclusion Criteria: Patients with systemic neoplasia, HIV, CKD or nephropathy from other etiologies, severe psychiatric disorders and pregnant women. Study design: This study consists of a randomized, cross-over, open-label controlled clinical trial. Patients will be randomly divided into two groups: GROUP 1 - insulin analog glargine once a day and GROUP 2 - NPH human insulin, three applications per day, both group will be treated with insulin lispro at mealtime. The laboratory tests will be performed at baseline and 12, 24, 36 and 48 weeks after the study start. During routine medical appointments will be analyzed self- monitoring of capillary blood glucose (SMBG) and the hypoglycemia score. After 24 weeks the basal insulin will be changed, i.e. patients using NPH insulin will receive insulin glargine and patients on insulin glargine will be changed to NPH insulin. A CGMS will be carried out at 24 and 48 weeks. Methodology: The metabolic profile will be evaluated throughout SMBG; biochemical, hormonal and hematological measurements; hypoglycemia score and CGMS. Statistical analysis will be performed using comparative descriptive analyzes, such as chi-square distribution, t-test and non-parametric tests. Analyze of data CGMS will include the area under the curve and the related statistic. Finally, logistic regression models will be adopted to evaluate the effect of the treatment on the several variables in question.

DETAILED DESCRIPTION:
This study consists of a randomized, cross-over, open-label controlled clinical trial. Randomized patients will be allocated alternately into two groups to receive the following therapies: GROUP 1 - insulin analog glargine once a day associated to insulin lispro at mealtime and GROUP 2 - NPH human insulin, three applications per day ( breakfast, lunch and bedtime) and insulin lispro at mealtime. Patients receiving insulin NPH plus insulin lispro will be oriented to mix both of them in the same syringe at breakfast and lunchtime. The laboratory tests will be performed at baseline and 12, 24, 36 and 48 weeks after the study start. During routine medical appointments the patient should bring the self- monitoring of capillary blood glucose (SMBG), eight points per day once a week, and hypoglycemia score.

After 24 weeks of insulin therapy, a continuous glucose monitoring system (CGMS) will be implemented for three days, and after that, the basal insulin changed i.e. patients using NPH insulin will receive insulin glargine and patients on insulin glargine will be changed to NPH insulin, both groups will keep insulin lispro before meals. A new CGMS will be carried out 24 weeks after therapy has been changed. Methodology: The metabolic profile will be evaluated throughout SMBG; biochemical, hormonal and hematological measurements; hypoglycemia score and CGMS (Medtronic/Northridge, CA). All randomized patients who use at least one dose of any study treatment will be considered in the Intent-to-treat (ITT) population. The initial plan is to randomize 40 patients, assuming a drop-out rate of 15%, to obtain a sample size of at least 34 randomized patients. .Statistical analysis will be performed using comparative descriptive analyzes, such as chi-square distribution, t-test and non-parametric tests. Analyze of data CGMS will include the area under the curve and the related statistic. Finally, logistic regression models will be adopted to evaluate the effect of the treatment on the several variables in question.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus and chronic kidney disease secondary to diabetic nephropathy in stages 3 and 4 (moderate and severe nephropathy, corresponding to glomerular filtration rate of 15-59 ml/min/1.73m²) will be included in the study.

Exclusion Criteria:

* Patients with systemic neoplasias,
* HIV, chronic kidney disease or nephropathy from other etiologies,
* severe psychiatric disorders
* pregnant women.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia S Queiroz, MD, PhD, Principal Investigator — Assistant Professor at Division of Endocrinology and Metabolism, Department of Internal Medicine, Clinic Hospital of the University of São Paulo Medical School
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Betonico CC, Titan SMO, Lira A, Pelaes TS, Correa-Giannella MLC, Nery M, Queiroz M. Insulin Glargine U100 Improved Glycemic Control and Reduced Nocturnal Hypoglycemia in Patients with Type 2 Diabetes Mellitus and Chronic Kidney Disease Stages 3 and 4. Clin Ther. 2019 Oct;41(10):2008-2020.e3. doi: 10.1016/j.clinthera.2019.07.011. Epub 2019 Aug 2. PMID 31383366

RESULTS

PARTICIPANT FLOW:
Groups:
- Glargine Insulin, Then NPH Insulin: The initial insulin dose for those randomized to IGlar was 80% of the total daily NPH dose that was being discontinued. All of them had pre-prandial Regular insulin switched to Lispro insulin (Humalog™, Lilly, Brazil), at the same dose as in use previously. After 24 weeks, basal insulins were switched; in other words, individuals on IGlar in the first period switched to INPH, and the doses of pre-meal insulin were sustained
- NPH Insulin, Then Glargine Insulin: The same total daily NPH insulin dose was maintained for those randomized to INPH. All of them had pre-prandial Regular insulin (Humulin R™, Lilly, Brazil) switched to Lispro insulin (Humalog™, Lilly, Brazil), at the same dose as in use previously. . After 24 weeks, basal insulins were switched; in other words, individuals on NPH in the first period switched to glargine insulin, and the doses of pre-meal insulin were sustained.
Period: First Intervention (24 Weeks)
Arm/Group | Glargine Insulin, Then NPH Insulin | NPH Insulin, Then Glargine Insulin
Started | 16 | 18
Completed | 14 | 15
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 2
Period: Second Intervention (24 Weeks)
Arm/Group | Glargine Insulin, Then NPH Insulin | NPH Insulin, Then Glargine Insulin
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine Insulin, Then NPH Insulin | NPH Insulin, Then Glargine Insulin | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (7.0) | 60.1 (8.7) | 61.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 18 | 34
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 19.0 (11.7) | 19.2 (7.0) | 19.1 (9.4)
Body weight [Mean (Standard Deviation); unit: kg] | 75.4 (11.9) | 82.6 (17.4) | 79.2 (15.3)
BMI [Mean (Standard Deviation); unit: kg/m²] | 28.6 (4.8) | 30.4 (4.3) | 29.6 (4.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 147 (22) | 136 (18) | 141 (20)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79 (12) | 75 (13) | 76 (12)

OUTCOME MEASURES:

1. Primary Outcome: Difference in A1c Levels
Description: A1c using high performance liquid chromatography measured in percentage
Time Frame: baseline and 24 weeks
Population: Primary endpoint A1c was assessed using an analysis of covariance (ANOVA) model.
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Glargine Insulin Period: This is an open-label, randomized, two-way crossover study, one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of insulin glargine, regardless of the sequence were grouped as glargine insulin.
- NPH Insulin Period: This is an open-label, randomized, two-way crossover study, one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of NPH insulin, regardless of the sequence were grouped as NPH insulin.
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 34 | 34
percentage
  Baseline | 8.86 (1.4) | 8.21 (1.3)
  24 weeks treatement | 7.95 (1.1) | 8.44 (1.3)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; A sample size of 34 participants (16 randomized to sequence IGlar/INPH and 18 randomized to sequence INPH/IGlar) provided 90% power to detect a mean difference of 0.7% in the primary endpoint (A1c), considering a 15% dropout rate and assuming an SD of 0.85%, and a type I error of 5%. Test for data normality (Kolmogorov-Smirnov statistics) was performed at baseline for each sequence of the therapy; Test type: Non-Inferiority or Equivalence — A sample size of 34 participants (16randomized to sequence IGlar/INPH and 18randomized to sequence INPH/IGlar) provided 90% power to detect a mean difference of 0.7% in the primary endpoint(A1c), considering a 15% dropout rate and assuming an SD of 0.85%, and a type I error of 5%; p = 0.00045, ANOVA — The intention-to-treat population consisted of all randomized participants

2. Primary Outcome: Number of Hypoglycemic Events
Description: Hypoglycemia was defined by capillary glycemia< 70 mg/dL (3.9 mmol/L), even if it was not accompanied by typical symptoms. Otherwise, hypoglycemia was classified as "severe" with SMBG below 50 mg/dL (2.8 mmol/L) or when it resulted in stupor, seizure, or unconsciousness that precluded self-treatment, thus requiring the assistance of another individual. Nocturnal events were defined as SMBG < 70mg/dL occurring after midnight and before wake-up in the morning (before 7:00am)12.
Time Frame: between 1rst and 24 weeks of each treatment arm
Population: Endpoint hypoglycemia was assessed using an analysis of covariance (ANOVA) model
Measure: Mean (Standard Deviation); unit: events per patients during 24 weeks
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 34 | 34
events per patients during 24 weeks
  total hypoglycemic events | 4.87 (5.39) | 6.34 (9.37)
  nocturnal hypoglycemias | 0.52 (1.03) | 1.52 (2.54)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; Analysis of covariance (ANOVA) model - total hypoglycemic events per patient during 24 weeks; Test type: Non-Inferiority or Equivalence — A sample size of 34 participants (16 randomized to sequence IGlar/INPH and 18 randomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%. Test for data normality (Kolmogorov-Smirnov statistics) was performed at baseline for each sequence of the therapy; p = 0.35, ANOVA — Analysis of covariance (ANOVA) model - total hypoglycemic events per patient during 24 weeks; number of total events per patient = 0 — The calculated value for the estimation parameter was zero, since the best treatment option for those with diabetes is reach a good glycemic control without hypoglycemia
Statistical Analysis 2: Comparison: Glargine Insulin Period vs NPH Insulin Period; A sample size of 34 participants (16randomized to sequence IGlar/INPH and 18 randomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%; Test type: Non-Inferiority or Equivalence — A sample size of 34 participants (16randomized to sequence IGlar/INPH and 18 randomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%; p = 0.047, ANOVA — Analysis of covariance (ANOVA) model - number of nocturnal hypoglycemic events per patient during 24 weeks; number of nocturnal events per patient = 0 — [estimate comment as in outcome 2, analysis 1]

3. Other Pre Specified Outcome: Glycemic Variability
Description: In order to observe variability in interstitial glucose levels related to the therapy in use, participants wore a blinded CGM for 3 days. Changes in glycemic patterns were expressed by the average daily time spent in hypoglycemia (≤70 mg/dL or <3.9 mmol/L), hyperglycemia (>180 mg/dL or >10 mmol/L) and euglycemia (70-180 mg/dL or 3.9-10 mmol/L).
Time Frame: 24 week
Population: Patients were excluded from the analysis because of unfamiliarity with mechanical procedures related to the CGM use, visual impairment or technical problems with the sensor measurement.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Glargine Insulin Period: This is an open-label, randomized, two-way crossover study, one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of NPH insulin, regardless of the sequence were grouped as glargine insulin.
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 24 | 24
percentage of time
  hyperglycemia | 30 (19) | 38 (19)
  normoglycemia | 67 (19) | 59 (19)
  hypoglycemia | 3 (6) | 3 (5)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; A sample size of 34 participants (16 randomized to sequence IGlar/INPH and 18 randomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%; Test type: Non-Inferiority or Equivalence — t-test was applied to compare percentages of the time spent in hypoglycemia, hyperglycemia and euglycemia on CGM readings; p < 0.05, t-test, 1 sided

4. Other Pre Specified Outcome: Total Daily Insulin Dose
Description: Daily total insulin dose at baseline compared to dose at week 24.
Time Frame: baseline and 24 weeks
Population: Randomization was stratified by the A1c value at baseline: <9.0% or ≥9.0%, in a 1:1 ratio, and the individuals who met all inclusion-criteria were allocated alternately to either an IGlar/INPH or an INPH/IGlar treatment sequence.
Measure: Mean (Standard Deviation); unit: units/Kg/day
Groups:
- Glargine Insulin: This is an open-label, randomized, two-way crossover study, one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of insulin glargine, regardless of the sequence were grouped as glargine insulin.
- NPH Insulin: This is an open-label, randomized, two-way crossover study, one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin. At the end of the study, all data acquired during the use of NPH insulin, regardless of the sequence were grouped as NPH insulin.
Arm/Group | Glargine Insulin | NPH Insulin
Number analyzed (Participants) | 34 | 34
units/Kg/day
  Baseline | 0.61 (0.21) | 0.63 (0.21)
  24 weeks treatment | 0.64 (0.26) | 0.64 (0.25)
Statistical Analysis 1: Comparison: Glargine Insulin vs NPH Insulin; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.668, ANOVA

5. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Time Frame: baseline and 24 weeks
Population: BMI endpoint was assessed using an analysis of covariance (ANOVA) model.
Measure: Mean (Standard Deviation); unit: Kg/m²
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 34 | 34
Kg/m²
  Baseline | 29.7 (4.7) | 30.0 (4.3)
  24 weeks treatement | 30.0 (4.3) | 30.4 (4.7)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; A sample size of 34 participants (16 randomized to sequence IGlar/INPH and 18r andomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%; Test type: Non-Inferiority or Equivalence — A sample size of 34 participants (16 randomized to sequence IGlar/INPH and 18r andomized to sequence INPH/IGlar) provided 90% power and assuming an SD of 0.85%, and a type I error of 5%; p = 0.999, ANOVA

6. Other Pre Specified Outcome: Serum Creatinine
Description: Creatinine is measured in milligrams per deciliter of blood (mg/dL
Time Frame: baseline and 24 weeks
Population: Creatinine endpoint was assessed using an analysis of covariance (ANOVA) model.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 34 | 34
mg/dL
  Baseline | 2.4 (0.7) | 2.5 (1.0)
  24 weeks treatement | 2.6 (0.8) | 2.6 (1.0)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.999, ANOVA

7. Other Pre Specified Outcome: Estimated Glomerular Filtration Rate (eGFR) Calculated by CKD-EPI
Description: Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation is one of the most widely used IDMS traceable equations for estimating GFR in patients age 18 and over. CKD-EPI equation includes variables for age, gender, and race, which may allow providers to observe that CKD is present despite a serum creatinine concentration that appears to fall within or just above the normal reference interval.
  CKD-EPI equation expressed as a single equation: GFR = 141 × min (Scr /κ, 1)α × max(Scr /κ, 1)-1.209 × 0.993Age × 1.018 [if female] × 1.159 [if black] where: Scr is serum creatinine in mg/dL, κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males,min indicates the minimum of Scr /κ or 1, and max indicates the maximum of Scr /κ or 1.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ml/min/1.7m²
Arm/Group | Glargine Insulin Period | NPH Insulin Period
Number analyzed (Participants) | 34 | 34
ml/min/1.7m²
  Baseline | 28.0 (9.6) | 27.4 (9.1)
  24 weeks treatement | 26.9 (10.0) | 25.9 (9.7)
Statistical Analysis 1: Comparison: Glargine Insulin Period vs NPH Insulin Period; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.994, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Description: hypoglycemia was classified as "severe" with SMBG below 50 mg/dL (2.8 mmol/L) or when it resulted in stupor, seizure, or unconsciousness that precluded self-treatment, thus requiring the assistance of another individual.
Groups:
- NPH Insulin: This is an open-label, randomized, two-way crossover study , one is IGlar/INPH treatment sequence and, another is INPH/IGlar sequence. Wherein, IGlar refers to glargine insulin and INPH refers to NPH insulin.
  At the end of the study, all data acquired during the use of NPH insulin, regardless of the sequence were grouped as NPH.
  NPH insulin: The same total daily NPH insulin dose was maintained for those randomized to INPH. All of them had pre-prandial Regular insulin (Humulin R™, Lilly, Brazil) switched to Lispro insulin (Humalog™, Lilly, Brazil), at the same dose as in use previously. . After 24 weeks, basal insulins were switched; in other words, individuals on NPH in the first period switched to glargine insulin, and the doses of pre-meal insulin were sustained.
Arm/Group | Glargine Insulin | NPH Insulin
Serious Adverse Events (participants affected / at risk) | 0/34 | 2/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine Insulin (N=34) | NPH Insulin (N=34)
Severe hypoglycemia (Nervous system disorders) | 0 (0) | 2 (2) — stupor, seizure, or unconsciousness that precluded self-treatment, thus requiring the assistance of another individual

LIMITATIONS AND CAVEATS:
The results only apply to patients with T2DM and DKD stages 3 and 4 and do not allow us to extrapolate any conclusion to those on dialysis or initial stages of DKD. The patients were randomized alternately, in accordance with the initial A1c.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No